CLINICAL TRIAL: NCT01954940
Title: THE EFFECT OF WHOLE BODY VIBRATION THERAPY UPON MUSCLE STRENGTH & FUNCTION IN AMBULATORY BOYS WITH DUCHENNE MUSCULAR DYSTROPHY
Brief Title: Whole Body Vibration Therapy in Boys With Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Dr. Leanne Ward, MD, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: # 12/17E
Record Dates: First submitted 2013-09-13; First posted 2013-10-07 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Whole body vibration therapy, muscle strength testing, bone health, ambulatory, endurance.
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Body Vibration Therapy (Experimental): Group will receive daily whole body vibration therapy for up to 9 minutes maximum at a maximum of 18 Hz.
  Interventions: Device: Whole Body Vibration Therapy
- Control group (No Intervention): Group will not receive whole body vibration therapy. This group will conduct all other tests and outcomes except whole body vibration therapy.

INTERVENTIONS:
Device: Whole Body Vibration Therapy
  Arms: Whole Body Vibration Therapy

SUMMARY:
Whole-body vibration therapy (WBVT) is a novel, non-pharmacological intervention aimed at improving muscle strength and endurance as well as bone density. It holds promise for children with neuromuscular disorders such as Duchenne muscular dystrophy (DMD) since muscle weakness results not only from muscle breakdown but also physical inactivity and muscle disuse atrophy. Weak DMD patients may increasingly limit their physical activity due to fear of falling or loss of independence (e.g. difficulty rising to stand without assistance). Prolonging the length of time boys with DMD are ambulatory is important for delaying complications of this disease (lung hypoventilation, scoliosis) as well as maintaining bone health. We propose to conduct a pilot study of WBVT in young boys with Duchenne muscular dystrophy (DMD). The primary outcome will be to document safety and feasibility of WBVT in this patient population. The secondary outcomes will evaluate changes in muscle strength and endurance. Bone health will also be examined as part of routine clinical care. The study will include 20 ambulatory boys with DMD; patients will be randomized (1:1 allocation) into 2 groups: WBVT treatment or no WBVT treatment (controls). Treatment groups will consist of 10 boys undergoing daily WBVT in an 8-week, open-label trial.

DETAILED DESCRIPTION:
Post-Study Completion Note: Given competition for enrollment in other DMD trials and burden from daily home WBVT training, it was not feasible to study WBVT in the trial setting, nor is it likely to be a feasible modality for optimizing musculoskeletal health in routine care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Duchenne muscular dystrophy confirmed by at least one of the following:

   * Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical presentation consistent with typical DMD
   * Positive gene deletion test (missing one or more exons) in the central rod domain (exons 25-60) of dystrophin, where reading frame can be predicted as "out-of-frame", and clinical presentation consistent with typical DMD
   * Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, or other mutation resulting in a stop codon mutation) definitively associated with DMD, and clinical presentation consistent with typical DMD
2. Age between 5 - 14 yrs old (inclusive)
3. Positive Gower sign (indicating ability to rise from the floor & presence of proximal muscle weakness).
4. Able to walk 10 meters in <12 seconds
5. Able to stand upon WBVT plate (with knees flexed) for entire treatment protocol (i.e. 15-minutes)
6. Stable absolute dose of glucocorticoids (i.e. prednisone or deflazacort) for at least 3 months prior
7. Stable absolute doses of all medication that may affect muscle function (i.e. coenzyme Q10, green tea extract, creatine, arginine, glutamine, nutritional supplements, etc.) for at least 3 months prior
8. Stable absolute dose of all medication that may affect bone metabolism (i.e. vitamin D and calcium supplementation) for at least 3 months prior

Exclusion Criteria:

1. Clinical presentation, genetic testing and/or muscle biopsy consistent with Becker muscular dystrophy
2. History of recent surgery (within past 6-months)
3. History of a recent fracture (long-bone or vertebral) within past 6-months.
4. Acute inflammatory processes of lower extremities (e.g. cellulitis, etc) due to risk of pain and/or worsening inflammatory process
5. History of venous thrombosis (theoretically risk of inducing thromboembolic event).
6. History of kidney or bladder stones
7. History of uncontrolled seizures or severe migraines
8. History of cardiac arrhythmia
9. Intracranial pathology or hardware (e.g. ventriculoperitoneal shunt, cochlear implant).
10. Use of any investigational or experimental products within last 6-months and/or concomitant participation in another study
11. Inability or refusal to follow the study requirements (e.g. autism, severe cognitive or behaviour problems)
12. Inability or refusal to provide informed consent (parent) and/or assent (child)

Ages: 8 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Assess the safety of using whole body vibration therapy in boys with Duchenne muscular dystrophy. To assess whether whole body vibration therapy can improve muscle strength and prolong ambulation from baseline to 8 weeks of therapy. To asses. | 8 weeks
  Is WBVT safe, convenient and well-tolerated when administered daily to ambulatory to boys with DMD?

SECONDARY OUTCOMES:
Does WBVT result in any change in muscle strength. | 8 weeks
  Does WBVT results in any measurable change in muscle strength measured by the maximum resistance of deltoid, hip flexor and knee extensor (measured with microFET2 dynamometer) and grip strength (measured by Jamar hand-held dynamometer)
Does WBVT result in any muscle function change. | 8 weeks
  Does WBVT results in any measurable change in muscle function as measured by timed functional testing (timed 10m walk test; timed 4-stair climb; timed Gower manoeuvre, 6-minute walk test)?
Does WBVT result in any measurable change in muscle endurance. | 8 weeks
  Does WBVT result in any measurable change in muscle endurance (total number of steps taken each day, measured by pedometer)?
Quality of life changes. | 8 weeks
  Does WBVT result in any change in patient and family reported quality of life report? Measured by the Peds Q of L questionnaire.
Gait changes. | 8 weeks
  Does WBVT result in any change in patient's gait (as measured by Gangway gait analysis and Leonardo force plate analysis)
Bone health | 8 weeks
  Does WBVT result in any change in bone health indices (as measured by pQCT and routine skeletal imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Ward, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada